CLINICAL TRIAL: NCT00104429
Title: A PhaseIIb, 96 Week, Randomised, Partially Double-blinded, Multicentre, Parallel Group, Repeat Dose Study to Evaluate the Safety, Tolerability, PK and Antiviral Effect of GW873140 in Combination With COMBIVIR (Lamivudine and Zidovudine) Upon Selected Immunological and Virological Markers of HIV-1 Infection in Antiretroviral Therapy Naive Adults
Brief Title: GW873140 In Combination With Combivir In HIV Infected Subjects
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102881
Record Dates: First submitted 2005-02-28; First posted 2005-03-01 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Infection, Human Immunodeficiency Virus I; HIV Infection
Keywords: HIV infections; therapy naive
MeSH Terms: conditions — Infections; HIV Infections | interventions — aplaviroc; lamivudine, zidovudine drug combination

INTERVENTIONS:
Drug: GW873140
Drug: Combivir
  Other Names: GW873140

SUMMARY:
This study is a 96-week study designed to evaluate the safety and efficacy of GW873140 in combination with Combivir in HIV infected, untreated subjects.

DETAILED DESCRIPTION:
A Phase IIb, 96 week, randomized, partially double-blinded, multicenter, parallel group, repeat dose study to evaluate the safety, tolerability, pharmacokinetics and antiviral effect of GW873140 in combination with Combivir (lamivudine and zidovudine) upon selected immunological and virological markers of HIV-1 infection in antiretroviral therapy naive adults

ELIGIBILITY:
Inclusion criteria:

* HIV infected subjects.
* Females must be of either non-childbearing age, or have a negative pregnancy test.
* All subjects participating in this study should be counseled on the practice of safe sex using a proven double barrier method of contraception throughout the study.
* Screening lab result of plasma HIV-1 RNA greater than or equal to 10,000 copies/mL and CD4 cell count greater than or equal to 100 cells/mm3.
* Have CC Chemokine Receptor5-tropic (R5-tropic) virus based on viral tropism test at screening visit.
* Have no drug resistance mutations in HIV-1 Reverse Transcriptase based on resistance test at screening visit.
* Be treatment-naive, defined as less than or equal to 2 weeks of treatment with a protease inhibitor (PI) or a nucleoside reverse transcriptase inhibitor/nucleotide reverse transcriptase inhibitor (NRTI/ NtRTI), or less than or equal to 7 days of therapy with a non-nucleoside reverse transcriptase inhibitor (NNRTI).
* Prior treatment with any entry inhibitor, attachment inhibitor, or fusion inhibitor (experimental or approved) is not allowed.
* Be able to understand and follow with protocol requirements, instructions and protocol-stated restrictions.
* Signed and dated written informed consent prior to study entry.

Exclusion criteria:

* Detection of any CXC Receptor4-tropic (X4-tropic) virus, based on viral tropism test at screening.
* Any drug resistance mutations in HIV-1 Reverse Transcriptase based on resistance test at screening visit.
* Active Class C AIDS-defining illness.
* Laboratory abnormalities at screen.
* Significant blood loss prior to study start.
* Pregnant or breastfeeding women.
* Additional qualifying criteria to be determined by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125
Dates: Start 2005-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with viral loads <400 copies/mL remaining on randomized treatment through Week 12

SECONDARY OUTCOMES:
- Comparison of safety and tolerability of different dosage regimens of GW873140 plus Combivir to standard of care regimen. - Assessment of drug resistance over time. - Co-receptor tropism following virological failure.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, MD, Study Director — GlaxoSmithKline
Locations (45):
- United States (24):
  - GSK Investigational Site, Bakersfield, California
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Stanford, California
  - GSK Investigational Site, Tarzana, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Vero Beach, Florida
  - GSK Investigational Site, Conyers, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Minneapolis, Minnesota
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Newark, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Providence, Rhode Island
  - GSK Investigational Site, Dallas, Texas
- GSK Investigational Site, Brussels, Belgium
- Canada (3):
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (4):
  - GSK Investigational Site, Levallois-Perret
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Nantes
  - GSK Investigational Site, Paris
- Germany (3):
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
- Italy (2):
  - GSK Investigational Site, Brescia, Lombardy
  - GSK Investigational Site, Milan, Lombardy
- Portugal (3):
  - GSK Investigational Site, Coimbra
  - GSK Investigational Site, Lisbon
  - GSK Investigational Site, Porto
- GSK Investigational Site, Madrid, Spain
- United Kingdom (4):
  - GSK Investigational Site, Manchester, Lancashire
  - GSK Investigational Site, Brighton, Sussex East
  - GSK Investigational Site, Birmingham, Warwickshire
  - GSK Investigational Site, London